CLINICAL TRIAL: NCT01913015
Title: An Open-Label, Phase I, Randomized Pharmacokinetic Study of Dietary Effects on Abiraterone Acetate Drug Levels in Patients With Metastatic Castration-Resistant Prostate Cancer (DEAL)
Brief Title: Dietary Fat Levels and Abiraterone Acetate Uptake in Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After enrollment of the first 3 subjects, an interim assessment was conducted. Comparing DBS sampling to plasma PK levels yielded unconvincing results.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9130; NCI-2013-01223 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA069533 (NIH)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (abiraterone acetate, low then high fat breakfast) (Experimental): Patients receive standard dose abiraterone acetate PO QD (held on days 2, 3, 9, and 10), and low-dose abiraterone acetate PO QD on days 3 and 10. Patients eat a low fat breakfast on day 3 and a high fat breakfast on day 10.
  Interventions: Drug: abiraterone acetate; Dietary Supplement: dietary intervention; Other: pharmacological study; Other: questionnaire administration; Other: laboratory biomarker analysis
- Arm II (abiraterone acetate, high then low fat breakfast) (Experimental): Patients receive abiraterone acetate as in Arm I. Patients eat a high fat breakfast on day 3, and a low fat breakfast on day 10.
  Interventions: Drug: abiraterone acetate; Dietary Supplement: dietary intervention; Other: pharmacological study; Other: questionnaire administration; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: abiraterone acetate — Given PO
  Other Names: CB7630; Zytiga
Dietary Supplement: dietary intervention — Receive low fat breakfast
  Other Names: Dietary Modification; intervention, dietary
Dietary Supplement: dietary intervention — Receive high fat breakfast
  Other Names: Dietary Modification; intervention, dietary
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: questionnaire administration — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized pilot phase I trial studies the side effects of dietary fat levels and abiraterone acetate uptake in patients with metastatic hormone-resistant prostate cancer. Abiraterone acetate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Eating a low or high fat diet may increase the uptake of abiraterone acetate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the dietary effects of a low fat and high fat diet at a low abiraterone acetate dose (250 mg) on drug levels compared to standard dose administered in a fasting condition.

SECONDARY OBJECTIVES:

I. To potentially guide decisions in the future to use low dose abiraterone in a fed state and decrease overall cost.

II. To evaluate the potential relationship between esterase activity and abiraterone metabolism in an exploratory analysis.

III. To determine the feasibility of using patient-collected dried blood spot (DBS) samples for pharmacokinetic monitoring.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive standard dose abiraterone acetate orally (PO) once daily (QD) (held on days 2, 3, 9, and 10), and low-dose abiraterone acetate PO QD on days 3 and 10. Patients eat a low fat breakfast on day 3 and a high fat breakfast on day 10.

ARM II: Patients receive abiraterone acetate as in Arm I. Patients eat a high fat breakfast on day 3, and a low fat breakfast on day 10.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* About to initiate or currently being treated with abiraterone acetate 1000 mg orally once daily
* Clinically able to receive abiraterone acetate in the opinion of the investigator in accordance with standard prescribing practices
* Ability to consume a low fat and high fat diet
* Expected duration of continuous abiraterone therapy > 8 weeks
* Signed and dated informed consent

Exclusion Criteria:

* Patients taking medications that strongly inhibit or induce cytochrome P450 (CYP)3A4 within 28 days prior to the start of the study will be excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC)0-24 measurement | Up to 24 hours (day 1)
  The cross-over difference (log[AUC0-24(low fat)] - log[AUC0-24(high fat)]) of each patient will be computed and graphically illustrated. The cross-over difference will be estimated and reported with 95% confidence interval. Hills-Armitage approach will be used to adjust for the period effect for the estimation. In addition, a bioequivalence range will be computed for the log(AUC0-24[1000 mg with fasting food]), allowing for 20% differences in each side.

SECONDARY OUTCOMES:
Accuracy of patient-collected DBS sampling technique | Day 3
  The first three patients enrolled will have duplicate venous blood samples obtained in clinic 2 hours post-dose for in vivo confirmation of the DBS methodology.
Patient adherence to pre-defined sampling schedule | Up to day 14
  Patients will document the date/time of drug administration and the date/time of sample collection using a drug and DBS sample diary. Deviations greater than 10% of the shorter of the two time intervals surrounding the pre-defined time point will be considered non-adherent. Adherence rates will be compared for different time points.
Patient satisfaction of DBS method, measured using the Patient Questionnaire of DBS Sampling Method | Day 14
  Paired t-test will be conducted to compare the DBC (or transformed DBC) for the evaluation of carry-over effect.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Beer, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States